CLINICAL TRIAL: NCT02711657
Title: Fibrocytes in Rheumatoid Arthritis, Asthma and Interstitial Lung-disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Søren Andreas Just, MD, Ph.D. Student, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S-20150172
Record Dates: First submitted 2016-03-13; First posted 2016-03-17 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Interstitial Lung Diseases; Rheumatoid Arthritis; Asthma
Keywords: Fibrocytes; Interstitial Lung Diseases; Rheumatoid Arthritis; Asthma
MeSH Terms: conditions — Lung Diseases, Interstitial; Arthritis, Rheumatoid; Asthma | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibrocyte measurement and lung function test (Experimental): All participants has a peripheral blood sample taken, where fibrocytes are measured using flowcytometry. Further peripheral blood mononuclear cells (PBMC) are isolated and cultured. All, except healthy controls, have their lung function measured.
  Interventions: Other: Fibrocyte measurement and lung function test.

INTERVENTIONS:
Other: Fibrocyte measurement and lung function test.

SUMMARY:
To study Fibrocytes in patients with Rheumatoid Arthritis, Interstitial lung disease and severe asthma and healthy controls.

DETAILED DESCRIPTION:
Objectives: 1) To demonstrate that circulating CD45+ CD34+ CD11b+ cells can express Procollagen 1 and thereby show that these markers can be used to identify circulating fibrocytes. 2) To measure the levels of circulating CD45+, CD34+, CD11b+ cells in patients with RA, Fibrotic ILDs, severe asthma and in healthy controls (HC). 3) To compare the levels with number of peripheral blood mononuclear cells (PBMC) that differentiate to mature fibrocytes in vitro.

Method: The CD45+, CD34+, CD11b+ cells from 4 patients were isolated by cell sorting, and stained for Procollagen. 30 patients (10 of each RA, fibrotic ILDs: IPF or non-specific interstitial pneumonitis (NSIP), severe asthma) and 10 HC were included. Current medication, disease activity, lung function and radiographic data were collected. In 100 µL of lysed blood cells were enumerated by flowcytometry. Further, PBMC were isolated and cultured for 5 days. Coverslips from two wells were stained and mature fibrocytes counted and reported as fibrocytes per 106 PBMC originally added to the well.

ELIGIBILITY:
Inclusion Criteria:

* 10 patient with rheumatoid arthritis.
* 10 patient with rheumatoid arthritis and interstitial lung disease
* 10 patients with interstitial lung disease (idiopathic pulmonary fibrosis or nonspecific interstitial pneumonia)
* 10 patients with asthma
* 10 healthy volunteers

Exclusion Criteria:

* Unable to sign written informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Measure fibrocytes in peripheral blood. | Baseline
  To measure the levels of circulating CD45+, CD34+, CD11b+ cells (cells/uL) in patients with RA, Fibrotic ILDs, severe asthma and in healthy controls (HC).

SECONDARY OUTCOMES:
Compare circulating CD45+, CD34+, CD11b+ cells (cells/uL) with number of fibrocytes in cultured cells (fibrocytes/cultured peripheral blood mononuclear cells). | Baseline
  To compare the levels of circulating CD45+, CD34+, CD11b+ cells (cells/uL) with number of peripheral blood mononuclear cells (PBMC) that differentiate to mature fibrocytes in vitro.
Fibrocytes and lung diffusion capacity. | Baseline
  Is the level of fibrocytes in peripheral blood (cells/uL) correlated signs of interstitial lung disease in a lung function measured by diffusing capacity for carbon monoxide (DLCO) (mmol CO per min per kPa).
Fibrocytes and rheumatoid arthritis | Baseline
  Is the level of fibrocytes in peripheral blood (cells/uL) correlated to disease activity in rheumatoid arthritis, measured by disease activity score in 28 joints (DAS28).

CONTACTS AND LOCATIONS:
Overall Officials: Søren Andreas Just, MD, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Just SA, Lindegaard H, Hejbol EK, Davidsen JR, Bjerring N, Hansen SWK, Schroder HD, Hansen IMJ, Barington T, Nielsen C. Fibrocyte measurement in peripheral blood correlates with number of cultured mature fibrocytes in vitro and is a potential biomarker for interstitial lung disease in Rheumatoid Arthritis. Respir Res. 2017 Jul 18;18(1):141. doi: 10.1186/s12931-017-0623-9. PMID 28720095